CLINICAL TRIAL: NCT06143488
Title: Endovascular Therapy Versus Best Medical Treatment for Acute Large Vessel Occlusion Stroke With Low NIHSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Wannan Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023090
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Acute Ischemic Stroke; Mild Neurocognitive Disorder; Thrombectomy
MeSH Terms: conditions — Ischemic Stroke; Neurocognitive Disorders

STUDY DESIGN:
Intervention Model Description: Drug: Best medical management Procedure: Endovascular therapy
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EVT group (Experimental): In the procedure, the methods including mechanical thrombectomy, aspiration thrombectomy, intra-arterial thrombolysis, angioplasty and stenting can be used according to the local interventionalists' choice.
  Interventions: Procedure: Endovascular therapy
- Best medical management (Active Comparator): All the patients enrolled received standard guideline-directed medical therapy including: monitor vital signs, management of blood pressure, glucose and lipids, antithrombotic (antiplatelet or anticoagulant therapy determined by treating physician) therapy if appropriate.
  Interventions: Procedure: Endovascular therapy; Drug: Best medical management

INTERVENTIONS:
Procedure: Endovascular therapy — Drug: Best medical management All the patients enrolled received standard guideline-directed medical therapy including: monitor vital signs, management of blood pressure, glucose and lipids, antithrombotic (antiplatelet or anticoagulant therapy determined by treating physician) therapy if appropriate.
  Procedure: Endovascular therapy In the procedure, the methods including mechanical thrombectomy, aspiration thrombectomy, intra-arterial thrombolysis, angioplasty and stenting can be used according to the local interventionalists' choice. Mechanical thrombectomy or aspiration thrombectomy will be recommended as the primary treatment.
Drug: Best medical management — All the patients enrolled received standard guideline-directed medical therapy including: monitor vital signs, management of blood pressure, glucose and lipids, antithrombotic (antiplatelet or anticoagulant therapy determined by treating physician) therapy if appropriate.
  Arms: Best medical management

SUMMARY:
Patients presenting with mild symptoms of acute ischemic stroke are common and account for approximately half of all acute ischemic stroke. About 30% of patients with minor stroke have a 90-day functional disability. Radiologically proven a large vessel occlusion (LVO) in patients with minor stroke is a well-established predictor of poor outcomes, while the poor outcomes following best medical management in patients with minor stroke with the underlying presence of a LVO are mainly driven by the occurrence of early neurological deterioration (END).

Considering the well-known strong association between lack of arterial recanalization and END, endovascular therapy (EVT) appears as an attractive option to improve functional outcomes for LVO-related patients with stroke with mild symptoms. Whether EVT is safe and effective in patients with mild stroke with an LVO is currently debated, since these patients were typically excluded from the pivotal EVT trials.

The current study aimed to further test the hypothesis that endovascular therapy would be superior to medical management with respect to functional recovery among low NIHSS patients caused by acute large-vessel occlusion in the anterior circulation.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years
* 2. Randomization can be finished within 24 hours from stroke onset (stroke onset time is defined as last known well time)
* 3.NIHSS score 2-5 at the time of randomization, but must include one of the following: any consciousness disorder (≥1 on NIHSS Question #1a); partial facial paralysis (≥1 on NIHSS Question #4); any weakness limiting sustained effort against gravity (≥1 on NIHSS Question #6 or #7); severe aphasia (≥1 on NIHSS Question #9), or visual or sensory extinction (≥1 on NIHSS Question #11).
* 4.CTA or MRA proven occlusion of the Internal Carotid Artery (ICA) terminal or M1/M2 segment of Middle Cerebral Artery
* 5.CTP/MRP Imaging shows the volume of Tmax>6s ≥ 50ml.
* 6. Informed consent signed

Exclusion Criteria:

* 1. Pre-stroke mRS score ≥1
* 2. Vascular occlusion caused by special causes is not suitable for endovascular treatment, such as Moyamoya disease, arteritis, radiation vascular disease, or fibromuscular development defective, and combined intracranial tumors, aneurysms, or intracranial arteriovenous malformations;
* 3. Severe comorbidities or unstable conditions, such as severe heart failure, pulmonary or renal failure (serum creatinine>2.8mg/dL or 250 µ mol/L or glomerular filtration rate <30ml/min), severe liver dysfunction and malignant tumors;
* 4. Any active bleeding or recent bleeding (gastrointestinal bleeding, urinary bleeding, etc.) in the past six months
* 5. Baseline platelet count <100×109 /L;
* 6. Refractory abnormal blood sugar that is difficult to control by medication (50mg/dL or 2.78mmol/L or 400mg/dL or 22.2mmol/L）;
* 7. Angiography shows a tortuous vascular pathway, making it difficult for the experimental equipment to reach the target position or retrieve it;
* 8. Known severe allergy for contrast agents or anesthetics;
* 9. Other circumstances that the investigator considers inappropriate for participation in the trial or that may pose significant risks to patients (such as inability to understand and/or follow the study procedures and/or follow up due to mental disorders, cognitive or emotional disorders)
* 10.The expected survival time is less than 1 year (such as patient with malignant tumor, advanced heart or lung diseases, etc.)
* 11.Participation in other interventional randomized clinical trials that may confound the outcome assessment of the trial;
* 12. Females who are pregnant, or those of childbearing, potential with positive urine or serum beta Human Chorionic Gonadotropin test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
90-day excellent clinical outcome | 90±7 days after randomization
  a dichotomized mRS 0-2 outcome

SECONDARY OUTCOMES:
Good clinical outcome | 90±7 days after randomization
  defined as a dichotomized mRS 0-2
early recovery | 72 hours after randomization
  72-hour NIHSS score≥4 points drop as compared with baseline

OTHER OUTCOMES:
Rate of symptomatic intracranial hemorrhage (sICH) per Heidelberg standard | within 72 hours after randomization
  Heidelberg standard was defined as new intracranial hemorrhage detected by brain imaging associated with any of the item below:
  4 points total NIHSS at the time of diagnosis compared to immediately before worsening.
  2 point in one NIHSS category. Leading to intubation/hemicraniectomy/ventricular drainage placement or other major medical/surgical intervention.
  Absence of alternative explanation for deterioration.
All-cause mortality rate | 90±7 days after randomization
  All-cause mortality rate

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Yijishan Hospital of Wannan Medical College, Wuhu, Anhui, China

IPD SHARING:
Plan to Share IPD: No